CLINICAL TRIAL: NCT00792025
Title: A Multicentre Phase II Trial to Determine the Efficacy of the Anti-Tyrosine Kinase Sunitinib (Sutent®) as Second Line Therapy in Patients With Transitional Cell Carcinoma (TCC) of the Urothelium Which Failed or Progressed After First Line Chemotherapy for Advanced or Metastatic Disease
Brief Title: Sunitinib as Second-Line Therapy in Treating Patients With Locally Advanced or Metastatic Transitional Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000618219; FRE-CRH-06-374-M; FRE CRH-VESSU; INCA-RECF0845; EUDRACT-2008-001004-22; PFIZER-FRE-CRH-06/374/M
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2009-07

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter
Keywords: metastatic transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; stage III bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; recurrent bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Sunitinib

INTERVENTIONS:
Drug: sunitinib malate

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying sunitinib to see how well it works as second-line therapy in treating patients with locally advanced or metastatic transitional cell cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the objective tumor response rate according to RECIST criteria in patients with locally advanced or metastatic transitional cell carcinoma of the urothelium treated with sunitinib malate who failed or progressed after first-line chemotherapy .

Secondary

* To determine the safety of this drug.
* To determine the time to response and duration of response.
* To determine the progression-free survival and overall survival of these patients.
* To evaluate the quality of life of these patients.

OUTLINE: This is a multicenter study.

Patients receive oral sunitinib malate once daily for 4 weeks. Courses repeat every 6 weeks for 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell cancer of the urothelium

  * Advanced or metastatic disease
  * Disease failed or progressed after first-line chemotherapy
* At least 1 non-irradiated measurable lesion assessed by CT scan or MRI according to RECIST
* No progressive brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (≤ 5 times ULN in presence of liver metastases)
* Creatinine clearance ≥ 40 mL/min
* PTT and INR ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during study treatment
* No uncontrolled high BP, defined as > 150/100 mm Hg despite treatment
* No diagnosis of a second malignancy within the past 5 years, except for basal cell or squamous cell carcinoma of the skin, incidental PT2 prostate cancer found on radical cystoprostatectomy material, or carcinoma in situ of the cervix, that has been adequately treated with no evidence of recurrence in the past 12 months
* None of the following within the past 12 months:

  * Myocardial infarction
  * Severe/unstable angina pectoris
  * Coronary artery bypass graft
  * Symptomatic congestive heart failure
  * Cerebrovascular accident
  * Transient ischemic attack
  * Pulmonary embolism
* At least 6 months since deep vein thrombosis
* No NCI CTCAE grade 3 hemorrhage within the past 4 weeks
* No pre-existing neuropathy ≥ NCI CTCAE grade 2
* No history of interstitial pneumonitis or pulmonary fibrosis
* No ongoing cardiac arrhythmias ≥ NCI CTCAE grade 2, atrial fibrillation of any grade, or prolongation of the QTc interval (> 450 msec for males or > 470 msec for females)
* No ongoing active infection
* No patients deprived of liberty or who are under supervision (including a trusteeship)
* No psychological, familial, sociological, or geographic condition potentially hampering compliance with study treatment and follow-up
* Patients must be affiliated to a social security system

PRIOR CONCURRENT THERAPY:

* Prior platinum-based therapy allowed
* No prior sunitinib malate
* No prior radiotherapy to ≥ 25% of marrow producing area
* Prior neoadjuvant or adjuvant chemotherapy allowed
* More than 2 weeks since prior and no concurrent oral anticoagulant agents at therapeutic doses

  * Low molecular weight heparin allowed
* At least 30 days since prior chemotherapy or radiotherapy and recovered
* No other concurrent anticancer treatment, including experimental agents, or participation in another investigational trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Objective response as assessed by RECIST criteria

SECONDARY OUTCOMES:
Progression-free survival
Overall survival
Time to response and duration of response
Safety
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Christine Theodore, MD, Principal Investigator — Hopital Foch
Locations (2):
- France (2):
  - Centre Rene Huguenin, Saint-Cloud
  - Hopital Foch, Suresnes